CLINICAL TRIAL: NCT07100379
Title: Balloon Inflation Time for Esophageal Strictures (BITES): A Randomized Multi-Center Study
Acronym: BITES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Jessica Lacy Yasuda, Attending Physician, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-P00048288
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Esophageal Atresia With Tracheo-esophageal Fistula; Esophageal Atresia; Esophageal Strictures
Keywords: endoscopic balloon dilation; post-surgical correction; esophageal strictures
MeSH Terms: conditions — Esophageal atresia with or without tracheoesophageal fistula; Esophageal Atresia; Esophageal Stenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (30 seconds) (Experimental): Patients who are randomized into Group A will undergo endoscopic balloon dilation for a total of 30 seconds.
  Interventions: Procedure: Endoscopic Balloon Dilation
- Group B (180 seconds) (Experimental): Patients randomized into Group B will undergo endoscopic balloon dilation for a duration of 180 seconds.
  Interventions: Procedure: Endoscopic Balloon Dilation

INTERVENTIONS:
Procedure: Endoscopic Balloon Dilation — Endoscopic balloon dilation is a routine procedure in which a catheter with a balloon is introduced into the esophagus to help treat esophageal strictures via endoscope. The catheter is placed directly across the span of the esophageal stricture and the balloon is inflated to pre-determined volume in order to dilate the esophageal stricture. Balloon will remain inflated for either 30 or 180 seconds based on patient's randomization.

SUMMARY:
Esophageal atresia (EA) is one of the most common gastrointestinal congenital anomalies that affects 1 in 2500 to 1 in 4000 live births. It is characterized by abnormal development of the esophagus, which requires surgical intervention to be compatible with life. Surgical repair of EA is associated with risk of developing esophageal strictures or narrowing, which nearly affects 40% of cases. Strictures can be treated using endoscopic balloon dilation, which consists of introducing a catheter with a balloon into the esophagus via endoscopy and positioning it across stricture followed by balloon inflation. The inflated balloon is held in position for a set amount of time with the goal to dilate the narrowed area. At this time there are no pediatric studies comparing difference balloon dilation times and outcomes. Our study's goal is to evaluate balloon dilation inflation time in treating esophageal anastomotic strictures to understand if inflation time is associated with outcome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with esophageal atresia with and without tracheoesophageal fistula, surgically repaired esophageal atresia, esophageal anastomotic strictures requiring endoscopic balloon dilation, and at least 1 endoscopic balloon dilation for esophageal anastomotic strictures within a 6 month period.

Exclusion Criteria:

* Patients who need endoscopic incisional therapy to manage anastomotic stricture during their first follow up endoscopy, patients requiring administration of intralesional steroid within 4 weeks of repair, have no follow up endoscopy within 6 months period, have any anastomosis type other than esophago-esophageal (e.g. jejunal or colonic interposition), and/or failure to meet target dilation time.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-06-24 (Estimated); Study Completion 2027-06-24 (Estimated)

PRIMARY OUTCOMES:
Stricture response to endoscopic balloon dilation | 6 months
  Study aims to determine whether the efficacy of endoscopic ballon dilation depends on duration of balloon inflation duration and does this influence the need for repeat endoscopic balloon dilations. Response to dilation will be defined by total number of dilations needed to treat stricture in a 6 month period.

SECONDARY OUTCOMES:
Change in esophageal anastomotic diameter | 6 months
  Secondary outcome measures will include esophageal anastomotic diameter at the conclusion of the study period compared to starting esophageal diameter.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Yasuda, MD, Principal Investigator — Boston Children's Hospital

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. Individual data will not provide us with an overall understanding of the efficacy of endoscopic ballon dilation, which is the primary goal of our study. This study will focus on analyzing the results obtained from the cohort as a whole and the results obtained from that analysis will be shared as part of a future manuscript.

REFERENCES:
- [Background] Khan AA, Shah SW, Alam A, Butt AK, Shafqat F, Castell DO. Pneumatic balloon dilation in achalasia: a prospective comparison of balloon distention time. Am J Gastroenterol. 1998 Jul;93(7):1064-7. doi: 10.1111/j.1572-0241.1998.00330.x. PMID 9672331
- [Background] Wallner O, Wallner B. Balloon dilation of benign esophageal rings or strictures: a randomized clinical trial comparing two different inflation times. Dis Esophagus. 2014 Feb-Mar;27(2):109-11. doi: 10.1111/dote.12080. Epub 2013 Apr 26. PMID 23621385
- [Background] Ten Kate CA, Tambucci R, Vlot J, Spaander MCW, Gottrand F, Wijnen RMH, Dall'Oglio L. An international survey on anastomotic stricture management after esophageal atresia repair: considerations and advisory statements. Surg Endosc. 2021 Jul;35(7):3653-3661. doi: 10.1007/s00464-020-07844-6. Epub 2020 Aug 3. PMID 32748272
- [Background] Kovesi T, Rubin S. Long-term complications of congenital esophageal atresia and/or tracheoesophageal fistula. Chest. 2004 Sep;126(3):915-25. doi: 10.1378/chest.126.3.915. PMID 15364774
- [Background] Castilloux J, Noble AJ, Faure C. Risk factors for short- and long-term morbidity in children with esophageal atresia. J Pediatr. 2010 May;156(5):755-60. doi: 10.1016/j.jpeds.2009.11.038. Epub 2010 Jan 31. PMID 20123142
- [Background] Serhal L, Gottrand F, Sfeir R, Guimber D, Devos P, Bonnevalle M, Storme L, Turck D, Michaud L. Anastomotic stricture after surgical repair of esophageal atresia: frequency, risk factors, and efficacy of esophageal bougie dilatations. J Pediatr Surg. 2010 Jul;45(7):1459-62. doi: 10.1016/j.jpedsurg.2009.11.002. PMID 20638524
- [Background] Krishnan U, Mousa H, Dall'Oglio L, Homaira N, Rosen R, Faure C, Gottrand F. ESPGHAN-NASPGHAN Guidelines for the Evaluation and Treatment of Gastrointestinal and Nutritional Complications in Children With Esophageal Atresia-Tracheoesophageal Fistula. J Pediatr Gastroenterol Nutr. 2016 Nov;63(5):550-570. doi: 10.1097/MPG.0000000000001401. PMID 27579697